CLINICAL TRIAL: NCT00342056
Title: Analysis of ABCG2 Genotype in Gleevec Treated Cancer Patients to Assess the Association of a Single Nucleotide Polymorphism (C421A) in ABCG2 and Response to Treatment
Brief Title: Role of Gene Variation in Effectiveness of Gleevec Treatment
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905090; 05-C-N090; NCT00897000 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2011-05

CONDITIONS: Cancer; Breast Cancer
Keywords: Pharmacogenetics; Transporter Proteins; Drug Exposure; Imatinib; Retrospective; Cancer
MeSH Terms: conditions — Neoplasms; Breast Neoplasms

SUMMARY:
This study will examine DNA from cancer patients previously treated with Gleevec to look for a variation (mutation) of the ABCG2 gene that may render the drug less effective in certain patients. Gleevec is used to treat chronic myeloid leukemia and gastrointestinal tumors. Although most patients respond to treatment, many with advanced disease develop resistance to the drug. It is thought that in some patients this resistance results from the action of a protein that causes Gleevec to be pumped out of the cells, reducing its usefulness.

Patients enrolled in clinical trials of Gleevec at the National Cancer Institute and at other participating institutions are eligible for this study.

DNA from patients' blood samples are analyzed for the ABCG2 gene and correlated with clinical data, such as the patient's age, race, disease state, weight, height, and body surface area. It will also look at the drug dose, how often the drug is given, the duration of treatment, side effects and other medications taken.

DETAILED DESCRIPTION:
ABCG2, also known as breast cancer resistance protein (BCRP), is an ATP-binding cassette (ABC) transporter that has been shown to confer resistance to several drugs, including mitoxantrone and topotecan. Gleevec (imatinib mesylate) has recently been identified as a substrate for ABCG2. The expression of ABCG2 in the human jejunum has been shown to be higher than expression MDR1, which encodes for P-glycoprotein. Therefore, it is plausible that the oral bioavailability of Gleevec could be dependent on the extent of transport. A single nucleotide polymorphism (C421A) has been identified in ABCG2 and has been shown in vitro to result in functional inactivation of this transporter protein. In this study, the relationship between the genotypes of ABCG2 and the pharmacokinetics or side effects will be retrospectively explored in patients with cancer who had been previously enrolled on clinical trials of Gleevec.

ELIGIBILITY:
* INCLUSION CRITERIA:

In this retrospective study, all cancer patients enrolled on IRB approved clinical trials of Gleevec from both the National Cancer and outside institutions will be eligible, provided that they have consented in the original consent form.

EXCLUSION CRITERIA:

Not applicable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-01; Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Washington Hospital Center, Washington D.C., District of Columbia, United States
- Katholieke Universiteit Leuven, U Hospitals UZ Gasthuisberg, Leuven, Belgium

REFERENCES:
- [Background] Bailey-Dell KJ, Hassel B, Doyle LA, Ross DD. Promoter characterization and genomic organization of the human breast cancer resistance protein (ATP-binding cassette transporter G2) gene. Biochim Biophys Acta. 2001 Sep 21;1520(3):234-41. doi: 10.1016/s0167-4781(01)00270-6. PMID 11566359
- [Background] Bates SE, Robey R, Miyake K, Rao K, Ross DD, Litman T. The role of half-transporters in multidrug resistance. J Bioenerg Biomembr. 2001 Dec;33(6):503-11. doi: 10.1023/a:1012879205914. PMID 11804192
- [Background] Leonard GD, Polgar O, Bates SE. ABC transporters and inhibitors: new targets, new agents. Curr Opin Investig Drugs. 2002 Nov;3(11):1652-9. PMID 12476969